CLINICAL TRIAL: NCT02835495
Title: The Healthy Living Partnerships to Prevent Diabetes in Veterans Pilot Study
Brief Title: Healthy Living Partnerships to Prevent Diabetes in Veterans Pilot Study
Acronym: HELP Vets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00033688; R34DK108100 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-18 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Pre-diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Weight Loss (Experimental): Behavioral: HELP Vets Intervention
  Lifestyle intervention consisting of 24 weekly group meetings led by a Veteran community health worker and 3 individual sessions with a nutritionist/diabetes educator
  Interventions: Behavioral: HELP Vets Intervention
- Enhanced Usual Care (Active Comparator): Behavioral: Individual Education Program
  Standard care consisting of 2 individual sessions with a nutritionist/diabetes educator and a monthly newsletter
  Interventions: Behavioral: Individual Education Program

INTERVENTIONS:
Behavioral: HELP Vets Intervention — This intervention involves a dietary weight loss program and an increase in caloric expenditure through moderate physical activity. The primary treatment objectives for the weight loss component of the intervention will be to decrease caloric intake in a nutritionally sound manner so as to produce a weight loss of approximately 0.3 kg per week for a total weight loss of 5-7%. The primary objective for the physical activity component of the intervention will be to promote an increase in home-based energy expenditure to an eventual goal of 180 min/week.
  Arms: Lifestyle Weight Loss
Behavioral: Individual Education Program — Participants will receive two individual sessions with a nutritionist during the first 3 months. In these sessions, the nutritionist will cover basic aspects of healthy eating and activity to support weight loss, discuss existing community resources and increased physical activity and weight loss. These participants will also receive a monthly newsletter on topics related to healthy lifestyle.
  Arms: Enhanced Usual Care

SUMMARY:
Diabetes and obesity are both major public health concerns and the prevalence of diabetes is even higher in the patient population of the Veterans Administration. This planning project is designed to adapt a successful weight-loss program for delivery through an existing outpatient clinic to reach local Veterans at risk for developing diabetes. The information gathered as a part of this project will be used to plan a larger trial designed to improve the health of Veterans by offering them a diabetes prevention program through their usual source of healthcare.

DETAILED DESCRIPTION:
Type II diabetes and its complications disproportionately affect the patient population served by the Department of Veterans Affairs (VA). Recent lifestyle interventions have demonstrated that weight-loss achieved through reductions in calorie intake and increases in physical activity can prevent or delay the onset of diabetes. The Healthy Living Partnerships to Prevent Diabetes (HELP PD), a community-based adaptation of the lifestyle intervention used in the Diabetes Prevention Program, achieved more than a 7% weight loss at 6 months.

In HELP Vets, researchers will test the feasibility of further translating the HELP PD lifestyle intervention, tailored for use in the Veteran population, in the Kernersville Community-Based Outpatient Clinic operated by the VA. The investigators plan to recruit 50 overweight or obese Veterans at high risk for developing diabetes from the existing patient population to participate in a 6-month weight loss intervention led by community health workers who are also Veterans. As VA outpatient clinics have the requisite infrastructure to identify, screen, and enroll participants and access to Veteran community health workers from within their patient populations, they are ideal potential homes for diabetes prevention programming. Data gathered during this planning grant will be used to develop a large-scale study to test implementing the HELP Vets intervention in a larger segment of the Veteran population.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-40 kg/m2
* Evidence of Pre-Diabetes: all participants will be required to qualify based on evidence of prediabetes from fasting plasma glucose, oral glucose tolerance test, or hemoglobin A1c (HbA1c) taken in the three months.
* The appropriate ranges for each test are
* Hemoglobin A1c (HbAlc): 5.7 to 6.4%
* Fasting Plasma Glucose: 95-125 mg/dL
* Oral Glucose Tolerance Test: 140-200 mg/dL.
* Blood measures will be collected from the medical record
* Prospective participants must be willing to accept randomization to either the lifestyle intervention or the enhanced usual care condition.

Exclusion Criteria:

* Currently involved in a supervised program for weight loss
* Clinical history of diabetes
* Clinical history of cardiovascular disease (CVD) occurring within the past 6 months, including myocardial infarction, angina, coronary revascularization, stroke, transient ischemic attack (TIA), carotid revascularization, peripheral arterial disease, and congestive heart failure
* Uncontrolled high blood pressure (BP > 160/100) Potential participants can be re-screened after controlled
* Pregnancy, planning pregnancy and breast feeding (self-report) during screening; Other chronic disease likely to limit lifespan to less than 2-3 years, including any cancer requiring treatment in past 5 years except non-melanoma skin cancer
* Chronic use of medicine known to significantly affect glucose metabolism (e.g., corticosteroids, protease inhibitors)
* Other conditions/criteria likely to interfere with participation and acceptance of randomized assignment, including the following: inability/unwillingness to give informed consent, another household member already randomized to HELP Vets, major psychiatric or cognitive problems (schizophrenia, dementia, self-reported active illegal substance or alcohol abuse), participation in another research study that would interfere with HELP Vets.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Z Vitolins, DrPH MPH RDN, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - W.G. "Bill" Hefner VA Medical Center, Salisbury, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 118 enrolled participants, 58 met inclusion criteria.
  51 participants were randomized. 1 had to withdraw pre-intervention initiation due to cancer diagnosis.
  50 participants were randomized and received the intervention treatment.
Groups:
- Lifestyle Weight Loss: Behavioral: HELP Vets Intervention
  Lifestyle intervention consisting of 24 weekly group meetings led by a Veteran community health worker and 3 individual sessions with a nutritionist/diabetes educator
  HELP Vets Intervention: This intervention involves a dietary weight loss program and an increase in caloric expenditure through moderate physical activity. The primary treatment objectives for the weight loss component of the intervention will be to decrease caloric intake in a nutritionally sound manner so as to produce a weight loss of approximately 0.3 kg per week for a total weight loss of 5-7%. The primary objective for the physical activity component of the intervention will be to promote an increase in home-based energy expenditure to an eventual goal of 180 min/week.
- Enhanced Usual Care: Behavioral: Individual Education Program
  Standard care consisting of 2 individual sessions with a nutritionist/diabetes educator and a monthly newsletter
  Individual Education Program: Participants will receive two individual sessions with a nutritionist during the first 3 months. In these sessions, the nutritionist will cover basic aspects of healthy eating and activity to support weight loss, discuss existing community resources and increased physical activity and weight loss. These participants will also receive a monthly newsletter on topics related to healthy lifestyle.
Period: Overall Study
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Started | 26 (26 randomized, however, one had to withdraw pre-intervention initiation due to cancer diagnosis.) | 25
Intervention Start | 25 | 25
Completed | 21 | 23
Not Completed | 5 | 2
Not completed — Cancer diagnosis prior intervention | 1 | 0
Not completed — Declined in-person follow-up visit | 4 | 2

BASELINE CHARACTERISTICS:
Population: 26 participants were randomized to the lifestyle weight loss intervention; however, one had to withdraw soon after randomization and before intervention initiation due to a cancer diagnosis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.5) | 64.2 (11.4) | 62.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 8 | 22
  White | 11 | 16 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51
Weight [Mean (Standard Deviation); unit: pounds] | 222.8 (32.6) | 231.9 (30.5) | 227.3 (31.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 133.5 (14.4) | 132.8 (12.4) | 133.2 (13.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81.0 (7.4) | 80.8 (7.5) | 80.9 (7.4)
Fasting Glucose [Count of Participants; unit: Participants] — In order to assess the feasibility of collecting this data from the electronic medical record, the proportion of participants for whom this data is available at randomization (+/- 90 days) will be reported.
  Participants | 18 | 24 | 42
Cholesterol (Lipid Panel) [Count of Participants; unit: Participants] — In order to assess the feasibility of collecting this data from the medical record, the proportion of participants for whom this data is available at randomization (+/- 90 days) will be reported.
  Participants | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Recruitment of Study Participants
Description: To characterize the ability to recruit Veterans to participate in this pilot study, the proportion of Veterans screened who are eligible to participate and the proportion of eligible participants who agree to participate will be calculated. The rate of referrals to the program by providers in the local community-based outpatient clinic will also be monitored.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Proportion of Eligible Participants of Total Screened: This reports the total number of participants who were screened and determined to be eligible for the study.
- Proportion of Eligible Participants Who Were Randomized: This reports the total number of participants who were randomized of those eligible for participation.
Arm/Group | Proportion of Eligible Participants of Total Screened | Proportion of Eligible Participants Who Were Randomized
Number analyzed (Participants) | 118 | 58
Participants | 58 | 51

2. Primary Outcome: Retention of Study Participants
Description: To characterize the ability to retain Veterans in this pilot study, the percentage of participants who complete the study (attendance at the 6-month assessment visit) as a measure of overall study retention will be calculated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25
Participants | 21 | 23

3. Primary Outcome: Adherence to the Lifestyle Weight Loss Intervention
Description: The proportion of intervention sessions attended will be calculated.
Time Frame: 6 months
Population: Participants in the Enhanced Usual Care Group were not asked to attend intervention sessions.
Measure: Mean (Inter-Quartile Range); unit: sessions attended
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 25 | 0
sessions attended | 14 [5 to 20] |

4. Other Pre Specified Outcome: Weight
Description: The means and standard deviations at 6 months will be calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 20 | 22
pounds | 210.4 (32.4) | 229.5 (34.5)

5. Other Pre Specified Outcome: Systolic Blood Pressure
Description: The means and standard deviations at 6 months will be calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 20 | 22
mmHg | 133.4 (14.1) | 133.8 (13.5)

6. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: The means and standard deviations at 6 months will be calculated.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 20 | 22
mmHg | 79.9 (11.6) | 82.3 (8.5)

7. Other Pre Specified Outcome: Proportion of Participants for Whom Fasting Glucose is Available at 6-months Post-randomization
Description: In order to assess the feasibility of collecting this data from the medical record, the proportion of participants for whom this data is available at 6-months post-randomization (+/- 90 days) will be reported.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25
Participants | 22 | 20

8. Other Pre Specified Outcome: Proportion of Participants for Whom Cholesterol (Lipid Panel) is Available at 6-months Post-randomization
Description: as for outcome 7
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25
Participants | 17 | 19

9. Other Pre Specified Outcome: Fasting Glucose
Description: The means and standard deviations at 6 months will be calculated.
Time Frame: 6 months
Population: Data not collected
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Cholesterol (Lipid Panel)
Description: The means and standard deviations at 6 months will be calculated.
Time Frame: 6 months
Population: Data not collected
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were reported at the 6-month follow-up visit using a standardized questionnaire.
Arm/Group | Lifestyle Weight Loss | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
As this was a pilot feasibility study, only a small number of participants were included and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT02835495/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT02835495/Prot_SAP_001.pdf